CLINICAL TRIAL: NCT06219811
Title: Prosthetic Maintenance Assessment for Two Implant-Retained Overdentures Reinforced With PEKK Versus Co-Cr Framework: A Randomized Controlled Clinical Trial
Brief Title: Prosthetic Maintenance of Two Implant-Retained Overdentures Reinforced With PEKK Versus Co-Cr Frameworks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M Refai, Lecturer of Oral and Maxillofacial Prosthodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec PC 122352
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Completely Edentulous
Keywords: Dental implants; Maintenance/standards; Overdenture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular implant-retained overdenture reinforced with a Co-Cr framework (Experimental): The patient received a mandibular implant-retained acrylic overdenture reinforced with a Co-Cr framework. The framework is manufactured by milling polymethylmethacrylate (PMMA) and then the PMMA undergo conventional casting to produce cobalt chromium (Co-Cr) framework. The framework included in the overdenture by conventional processing technique.
  Interventions: Device: Two implant -retained overdenture reinforced with Co-Cr framework
- Mandibular implant-retained overdenture reinforced with a PEKK framework (Active Comparator): The patient received a mandibular implant-retained acrylic overdenture reinforced with a Polyetherketoneketone (PEKK) framework. The framework is manufactured by milling PEKK the framework included in the overdenture by conventional processing technique.
  Interventions: Device: Two implant -retained overdenture reinforced with PEEK framework

INTERVENTIONS:
Device: Two implant -retained overdenture reinforced with Co-Cr framework — The intervention is made from polymethylmethacrylate reinforced with cobalt chromium ( Co-Cr) framework.
  Other Names: implant retained overdenture
  Arms: Mandibular implant-retained overdenture reinforced with a Co-Cr framework
Device: Two implant -retained overdenture reinforced with PEEK framework — The intervention is made from polymethylmethacrylate reinforced with Polyetherketoneketone ( PEEK) framework.
  Other Names: implant retained overdenture
  Arms: Mandibular implant-retained overdenture reinforced with a PEKK framework

SUMMARY:
The goal of this randomized clinical trial is to compare and assess the prosthetic maintenance of two implant-retained mandibular overdentures reinforced with PEKK and Co-Cr frameworks after twelve months. Twenty-four participants were randomly assigned to two groups: Group I received a mandibular implant-retained overdenture reinforced with a Co-Cr framework, while Group II received a mandibular implant-retained overdenture reinforced with a PEKK framework. Also, both groups were rehabilitated with a maxillary complete removable denture.

DETAILED DESCRIPTION:
Twenty-four participants with edentulous maxillary and mandibular ridges underwent meticulous selection, with two implants placed in the mandibular canine areas through a two-stage surgical technique facilitated by a radiographic and surgical stent. Following this, patients were provided with maxillary and mandibular complete removable dentures relined with soft liners. After the subsequent three-month osseointegration period, ball attachments were introduced. Patients were randomly allocated to two groups based on the type of prosthesis they received. Group I received mandibular implant-retained overdenture reinforced with the Co-Cr framework, while Group II received mandibular implant-retained overdenture reinforced with the PEKK framework, both groups received complete removable dentures for the maxillary arch. The assessment of prosthetic maintenance for mandibular implant-retained overdentures in both groups was conducted twelve months post-denture insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 50-70 years old.
* Completely edentulous patients
* Systemically free from any disease that contraindicates implant placement.
* A minimum of 12 -15 millimeters of bone height and 6 mm bone width at canine areas diagnosed from the pre-operative cone beam CT.
* Sufficient inter-arch space (15mm) to accommodate the mandibular implant-retained overdentures.

Exclusion Criteria:

* Patients with bone or mucosal diseases.
* Heavy smokers.
* Patients with uncontrolled metabolic disorders such as diabetes mellitus.
* Patients with parafunctional habits.
* Patients with conditions that might complicate the treatment, such as: severe gag reflex, limited mouth opening.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Prosthetic Maintenance of both types of implant retained overdentures | twelve months after delivery of implant retained overdenture
  Evaluation of prosthetic maintenance for mandibular implant-retained overdentures in both groups was made after twelve months of overdenture insertion. Prosthetic maintenance is a checklist for the following aspects that were inspected regarding screw (screw loosening, screw fracture), attachments (wear, distortion, fracture, replacement), and overdentures (reline, remake, fracture, teeth wear, teeth separation, or fracture).maintenance for complication assed through counting frequency of incidence. The unit of measurement used is percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Omnia MS Refai, PHD, Principal Investigator — Faculty of Dentistry ,Ain Shams University; Heba A Salama, PHD, Principal Investigator — Faculty of Dentistry , Misr International Univeristy
Locations (1):
- Faculty of Dentistry, Ain shams University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No